CLINICAL TRIAL: NCT04965285
Title: Operating Surgical Checklist Completion Out Before Surgical Procedures
Brief Title: Operating Room WHO Surgical Safety Checklist Process Completion: an Observational Study
Status: Completed | Type: Observational
Sponsor: Nepal Mediciti Hospital (Other)
Responsible Party: Principal Investigator, Bikash Khadka, Principal Investigator, Nepal Mediciti Hospital
Other Study IDs: 2589
Record Dates: First submitted 2021-06-30; First posted 2021-07-16 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Safety Issues; Patient Acceptance of Health Care
Keywords: Time Out, Healthcare
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: quality assesment — For each time-out procedure observed, the investigators will record compliance for each element of the time-out. Elements that are clearly verbalized by the member of the operating room team performing the time-out were considered compliant.
  As each step of the time-out is verbalized by a team member, the operating room team members are expected to respond. The observations will be conducted by trained study staff using a standardized Checklist/ Proforma to assess surgical team compliance with the time-out protocol and to record general observations of the operating room environment. Any non-routine events that occurred during the time-out process will be recorded.
  In each phase, the Checklist coordinator must be permitted to confirm that the team has completed its tasks before it proceeds onward.

SUMMARY:
The WHO Surgical Safety Checklist is a simple tool designed to improve the safety of surgical procedures by bringing together the whole operating team (surgeons, anaesthesia providers and nurses) to perform key safety checks during vital phases of perioperative care: prior to the induction of anesthesia, prior to skin incision and before the team leaves the operating room.

In 2007, WHO Patient Safety launched the Second Global Patient Safety Challenge, Safe Surgery Saves Lives.Anaesthetists, operating theatre nurses, surgeons, safety experts, patients and other professionals came together and came up with the WHO Surgical Safety Checklist. The 19 items of the surgical checklist have shown to improve on mortality and morbidity.

Surgical time out is carried out before the start of any surgical procedures to reduce the occurrence of wrong-site, wrong-procedure, and wrong-person surgery where the patient's identity, the procedure, and the surgical site before surgical incision or the start of the procedure is verified. This also helps to raise any concern regarding the procedural risk and any concerns, prevent medical errors, patient morbidity, patient mortality, and reduce surgical complication rates.

The Checklist is intended as a tool for use by clinicians interested in improving the safety of their operations and reducing unnecessary surgical deaths and complications and also help ensure that teams consistently follow a few critical safety steps and thereby minimize the most common and avoidable risks endangering the lives and wellbeing of surgical patients .

The aim of this Checklist is to reinforce accepted safety practices and foster better communication and teamwork between clinical disciplines.

DETAILED DESCRIPTION:
Definition of terms A time-out is defined as "an immediate pause by the entire surgical team to confirm the correct patient, procedure, and site," for Preventing Wrong Site, Wrong Procedure, and Wrong Person Surgery for all accredited hospitals, ambulatory care centers, and office-based surgery facilities Elements that are clearly verbalized by the member of the operating room team performing the time-out were considered compliant Distraction is defined as any involvement in an activity concerning a non-life-threatening issue by any operating room team member, including conversations unrelated to the time-out, loud music playing, unexpected entrances, and personnel engaged in other tasks, among others.

The Checklist divides the operation into three phases, each corresponding to a specific time period in the normal flow of a procedure-the period before induction of anaesthesia, the period after induction and before surgical incision, and the period during or immediately after wound closure but before removing the patient from the operating room.

For each time-out procedure observed, the investigators will record compliance for each element of the time-out. Elements that are clearly verbalized by the member of the operating room team performing the time-out were considered compliant.

As each step of the time-out is verbalized by a team member, the operating room team members are expected to respond. The observations will be conducted by trained study staff using a standardized Checklist/ Proforma to assess surgical team compliance with the time-out protocol and to record general observations of the operating room environment. Any non-routine events that occurred during the time-out process will be recorded.

In each phase, the Checklist coordinator must be permitted to confirm that the team has completed its tasks before it proceeds onward.

Anticipated and actual blood loss, anticipated and actual surgical duration will also be noted

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years surgical patients undergoing surgery at Nepal Mediciti Hospital

Exclusion Criteria:

* Emergency surgical cases, patients not being able to participate verbally

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: all surgical cases for elective surgeries, aged 18 and above, will be included on this study
Sampling Method: Non-Probability Sample
Enrollment: 322 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-28 (Actual)

PRIMARY OUTCOMES:
Quality of execution of the WHO surgical safety checklist in routine clinical practice | 1 day
  to evaluate for quality of execution of WHO surgical safety checklist during routine practice before every surgical procedures in our institute.

SECONDARY OUTCOMES:
To evaluate for any distractions and interruptions, deviations from protocol, and the problem-solving strategies used by operating room team members to mitigate the non routine events | 1 day
  to check for any factors that distracts or disturbs during conductance of WHO surgical checklist.
  to evaluate if there has been any deviation from protocol to check for any non routine events and any measures taken to overcome them

CONTACTS AND LOCATIONS:
Overall Officials: bikash khadka, MD, Principal Investigator — Nepal Mediciti Hospital
Locations (1):
- Nepal mediciti Hospital, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: Yes
research data will be made available if requested or contacted via Email services
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Actual Study Start Date: May 2021 Estimated Primary Completion Date: January 2022 Estimated Study Completion Date: February 2022
Access Criteria: On contact via Email services, description will be made available